CLINICAL TRIAL: NCT04057365
Title: A Single Arm Phase II Study of the Combination of DKN-01 and Nivolumab in Previously Treated Patients With Advanced Biliary Tract Cancer (BTC)
Brief Title: Study of the Combination of DKN-01 and Nivolumab in Previously Treated Patients With Advanced Biliary Tract Cancer (BTC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on a Simon 2-stage design, this study did not meet response criteria to proceed to stage 2.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry); Leap Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Joseph Franses, MD, PHD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-200
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Results first posted 2024-04-10 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Biliary Tract Cancer
Keywords: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DKN 01 and Nivolumab Safety Run in (Experimental): * DKN-01 will be administered intravenously on day 1 and day 15 of each 28 day cycle
  * Nivolumab will be administered intravenously on day 1 and day 15 of each 28 day cycle
  Interventions: Drug: Nivolumab; Drug: DKN-01
- DKN 01 and Nivolumab (Experimental): * DKN-01 will be administered intravenously on day 1 and day 15 of each 28 day cycle
  * Nivolumab will be administered intravenously on day 1 and day 15 of each 28 day cycle
  Interventions: Drug: Nivolumab; Drug: DKN-01

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is believed to work by attaching to and inhibiting a specific protein in the cancer that controls parts of the immune system (the system in the body that fights off infections and diseases) by shutting down certain immune responses. The investigators believe that nivolumab will inhibit the protein, thus allowing the immune cells to recognize and destroy cancer cells.
  Other Names: Opdivo
Drug: DKN-01 — DKN-01 is believed to work by attaching to and inhibiting (stopping) a specific pathway in the cells that is responsible for processes such as cell growth

SUMMARY:
This research is studying the effect of the combination of how two study drugs (Nivolumab and DKN-01) works in people with advanced biliary tract cancer.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The U.S. Food and Drug Administration (FDA) has not approved DKN-01 as a treatment for any disease.

The FDA has not approved nivolumab for this specific disease but it has been approved for other cancers.

DKN-01 and nivolumab are both antibodies. An antibody is a protein that attaches to other cells to fight off infection. DKN-01 is believed to work by attaching to and inhibiting (stopping) a specific pathway in the cells that is responsible for processes such as cell growth. Nivolumab is believed to work by attaching to and inhibiting a specific protein in the cancer that controls parts of the immune system (the system in the body that fights off infections and diseases) by shutting down certain immune responses. The investigators believe that nivolumab will inhibit the protein, thus allowing the immune cells to recognize and destroy cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed intra- or extrahepatic cholangiocarcinoma or gallbladder cancer
* Participants must have measurable disease by CT/MRI by RECIST version 1.1 criteria
* Prior chemoembolization, radiofrequency ablation, or radiation to the liver is allowed as long as the patient has measurable disease outside of the treated area or measurable progression per RECIST v1.1 at the site of the treated area.
* Documented progression after ≥1 line of systemic therapy for advanced BTC. Prior adjuvant chemotherapy qualifies as this 1 line if the last cycle of adjuvant therapy was completed within 6 months of radiological progression.
* Age ≥ 18 years
* ECOG performance status ≤1
* Life expectancy of greater than 3 months
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥1,500/mcL
  * Absolute lymphocyte count ≥1.0 x 10^9/L
  * Platelets ≥75,000/mcL
  * Hemoglobin ≥ 8.0 g/dL (prior transfusions are allowed if given ≥ 7 days before testing)
  * Total bilirubin < 2.0 x institutional upper limit of normal; except patients with Gilbert Syndrome who must have a total bilirubin level of < 3.0 x ULN
  * AST(SGOT)/ALT(SGPT) ≤3 × institutional upper limit of normal; < 5 x ULN in case of liver metastases
  * Creatinine < 2.0 x institutional upper limit of normal OR Creatinine clearance ≥30 mL/min/1.73 m2 for participants with creatinine levels ≥ ULN
  * International Normalized Ratio (INR) ≤ 1.5 x ULN unless patient is receiving anticoagulant therapy as long as INR is within therapeutic range of intended use of anticoagulants
  * Serum albumin > 2.5 g/dL
* Subjects with hepatitis B or C are eligible to enroll if they have:

  * Chronic HBV infection (evidenced by a positive HBV surface antigen or HBV DNA) as long as they have been on antiviral therapy for ≥ 4 weeks.
  * Chronic or resolved HCV infection (evidenced by a detectable HCV RNA or antibody). Antiviral therapy is not required for chronic HCV.
* Women of child-bearing potential and men must agree to use adequate contraception according to national guidelines (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 5 months for women and 7 months for men after completion of study drug administration.
* Female subjects must be either of non-reproductive potential (i.e., post-menopausal by history: ≥ 50 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior DKK1 inhibitor or anti-PD-1/PD-L1 treatment
* Participants with Child-Pugh B or C cirrhosis
* Participants with a diagnosis of ampullary cancer
* Treatment with any of the following within the specified time frame prior to the first dose of DKN-01 and nivolumab:

  * Any non-investigational or investigational anticancer therapy within 3 weeks or have not recovered from side effects of such therapy prior to treatment administration (mitomycin within prior 5 weeks). For targeted therapy, 5 half-lives are sufficient, even if <3 weeks. Concurrent participation in an observational study may be allowed after review by the Principal Investigator.
  * Patients with locoregional therapy, e.g., transarterial chemoembolization (TACE), selective internal radiotherapy (SIRT), external beam radiation, or ablation within 4 weeks
  * Palliative limited field radiotherapy (i.e. bone metastases) within 2 weeks
  * Major surgery within the previous 4 weeks (the surgical incision should be fully healed prior to the first dose of treatment)
* Fredericia's corrected QT interval (QTcF) ≥ 500 ms on ECG conducted during screening
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to DKN-01 or Nivolumab.
* A serious illness or medical condition(s) including, but not limited to, the following:

  * Known brain metastasis (not including primary brain tumors) unless patient is clinically stable for ≥ 1 month without systemic corticosteroids beyond physiologic replacement (>10 mg prednisone daily).
  * Known acute systemic infection.
  * Myocardial infarction, severe/unstable angina, symptomatic congestive heart failure
  * New York Heart Association [NYHA] Class III or IV (see Appendix D, New York Heart Association [NYHA] Classification) within the previous 2 months; if >2 months, cardiac function must be within normal limits and the patient must be free of cardiac-related symptoms.
  * Chronic nausea, vomiting, or diarrhea considered to be clinically significant in the opinion of the investigator.
  * Congenital long QT syndrome, or any known history of torsade de pointes, or family history of unexplained sudden death.
  * Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that in the judgment of the investigator would make the patient inappropriate for entry into this study.
* Patients with a history of another primary malignancy that is currently clinically significant, and has potential for metastases or currently requires active intervention (except for hormonal therapy for breast or prostate cancer).
* Any condition requiring systemic treatment with either corticosteroids (> 2mg daily dexamethasone equivalent) or other immunosuppressive medications within 14 days of starting the study medications. Premedication for hypersensitivity reactions (e.g. to contrast for CT or gadolinium for MRI) is allowed.
* Subjects with autoimmune disease active within the last two years including but not limited to Crohn's disease, ulcerative colitis, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, type I diabetes mellitus, vasculitis, or glomerulonephritis

  * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible for this study.
  * Patients with controlled Type I diabetes mellitus on a stable insulin regimen are eligible
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis/fibrosis in the radiation field is permitted.
* Patients who received treatment with live vaccines within 30 days prior to the first dose of study medication. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, shingles, yellow fever, seasonal flu, H1N1 flu, rabies, BCG and typhoid vaccine.
* History of osteonecrosis of the hip or evidence of structural bone abnormalities in the proximal femur on magnetic resonance imaging (MRI) scan that is symptomatic and clinically significant. Degenerative changes of the hip joint are not excluded.
* Known osteoblastic bony metastasis. Screening of asymptomatic subjects without a history of metastatic bony lesions is not required.
* Prior allogeneic stem cell or solid organ transplant.
* Known or current evidence of HIV
* Pregnant or lactating female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2022-09-25 (Actual); Study Completion 2022-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Franses, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: MGH - Contact the Partners Innovations team at http://www.partners.org/innovation
URL: http://www.partners.org/innovation

RESULTS

PARTICIPANT FLOW:
Groups:
- DKN 01 and Nivolumab Safety Run in; DKN 01 and Nivolumab: * DKN-01 will be administered intravenously on day 1 and day 15 of each 28 day cycle
  * Nivolumab will be administered intravenously on day 1 and day 15 of each 28 day cycle
  Nivolumab: Nivolumab is believed to work by attaching to and inhibiting a specific protein in the cancer that controls parts of the immune system (the system in the body that fights off infections and diseases) by shutting down certain immune responses. The investigators believe that nivolumab will inhibit the protein, thus allowing the immune cells to recognize and destroy cancer cells.
  DKN-01: DKN-01 is believed to work by attaching to and inhibiting (stopping) a specific pathway in the cells that is responsible for processes such as cell growth
Period: Overall Study
Arm/Group | DKN 01 and Nivolumab Safety Run in | DKN 01 and Nivolumab
Started | 15 | 0
Completed | 13 | 0
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: Based on a Simon 2-stage design, this study did not meet response criteria to proceed beyond the safety run-in group.
Groups:
- Total: Total of all reporting groups
Arm/Group | DKN 01 and Nivolumab Safety Run in | DKN 01 and Nivolumab | Total
Number analyzed (Participants) | 15 | 0 | 15
Age, Customized [Count of Participants; unit: Participants]
  18 - 65 years | 7 | 0 | 7
  >65 years | 8 | 0 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 0 | 6
  Male | 9 | 0 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 0 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response is evaluated using Response Evaluation Criteria in Solid Tumors criteria (RECIST 1.1). A participant is considered to have responded if they achieve either of the following outcomes:
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm
  * Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters
Time Frame: up to 1 year
Population: A Simon 2 stage design will be used, and the study did not meet criteria to proceed beyond the safety run-in cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | DKN 01 and Nivolumab Safety Run in | DKN 01 and Nivolumab
Number analyzed (Participants) | 13 | 0
Participants | 0 |

2. Secondary Outcome: Progression Free Survival
Description: Progression-Free Survival (PFS) is defined as the time from registration to the earlier of disease progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation.
  Disease progression is assessed using RECIST 1.1 criteria:
  - Progressive Disease(PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: up to 1 year
Population: A Simon 2 stage design will be used, and the study did not meet criteria to proceed beyond the safety run-in cohort.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | DKN 01 and Nivolumab Safety Run in | DKN 01 and Nivolumab
Number analyzed (Participants) | 13 | 0
days | 49 [40 to 96] |

3. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) is defined as the time from registration to death due to any cause, or censored at date last known alive.
Time Frame: up to 1 year
Population: A Simon 2 stage design will be used, and the study did not meet criteria to proceed beyond the safety run-in cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | DKN 01 and Nivolumab Safety Run in | DKN 01 and Nivolumab
Number analyzed (Participants) | 13 | 0
Participants | 12 |

4. Secondary Outcome: Treatment Emergent Adverse Events
Description: Treatment emergent adverse events (TEAEs) are undesirable events not present prior to study treatment, or an already present event that worsens either in intensity or frequency following the treatment. TEAEs reported below were assessed as grade 3 or higher according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v 5.0) guidelines.
Time Frame: up to 1 year
Population: The study did not proceed beyond the initial safety run-in cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | DKN 01 and Nivolumab Safety Run in | DKN 01 and Nivolumab
Number analyzed (Participants) | 13 | 0
Participants
  Abdominal pain | 2 |
  Lymphopenia | 2 |
  Alanine aminotransferase (ALT) increased | 1 |
  Aspartate aminotransferase (AST) increased | 1 |
  Alkaline phosphatase increased | 1 |
  Dyspnea | 1 |
  Hypokalemia | 1 |

ADVERSE EVENTS:
Time Frame: up to 1 year
Description: A Simon 2 stage design will be used, and the study did not meet criteria to proceed beyond the safety run-in cohort.
Arm/Group | DKN 01 and Nivolumab Safety Run in | DKN 01 and Nivolumab
All-Cause Mortality (participants affected / at risk) | 1/13 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/0
Other Adverse Events (participants affected / at risk) | 13/13 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DKN 01 and Nivolumab Safety Run in (N=13) | DKN 01 and Nivolumab (N=0)
Aspartate aminotransferase increased (Investigations) | 9 | NA
Anemia (Blood and lymphatic system disorders) | 7 | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | NA
Hyponatremia (Metabolism and nutrition disorders) | 7 | NA
Alanine aminotransferase increased (Investigations) | 6 | NA
Fatigue (General disorders) | 6 | NA
Abdominal pain (Gastrointestinal disorders) | 5 | NA
Alkaline phosphatase increased (Investigations) | 5 | NA
Anorexia (Gastrointestinal disorders) | 5 | NA
Ascites (Gastrointestinal disorders) | 5 | NA
Diarrhea (Gastrointestinal disorders) | 5 | NA
Lymphocyte count decreased (Investigations) | 5 | NA
Nausea (Gastrointestinal disorders) | 4 | NA
Blood bilirubin increased (Investigations) | 3 | NA
Fever (General disorders) | 3 | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | NA
Peripheral sensory neuropathy (Nervous system disorders) | 3 | NA
Platelet count decreased (Investigations) | 3 | NA
Pruritus (Skin and subcutaneous tissue disorders) | 3 | NA
Edema limbs (General disorders) | 3 | NA
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 2 | NA
Chills (General disorders) | 2 | NA
Constipation (Gastrointestinal disorders) | 2 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | NA
Dehydration (Metabolism and nutrition disorders) | 2 | NA
Dizziness (Nervous system disorders) | 2 | NA
Headache (Nervous system disorders) | 2 | NA
Hyperglycemia (Metabolism and nutrition disorders) | 2 | NA
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | NA
Neutrophil count decreased (Investigations) | 2 | NA
Pain (General disorders) | 2 | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | NA
Sinus tachycardia (Cardiac disorders) | 2 | NA
Lung infection (Infections and infestations) | 2 | NA
Abdominal distension (Gastrointestinal disorders) | 1 | NA
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | NA
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Atrial fibrillation (Cardiac disorders) | 1 | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | NA
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | NA — systolic murmur
Creatinine increased (Investigations) | 1 | NA
Death NOS (General disorders) | 1 | NA
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | NA
Duodenal ulcer (Gastrointestinal disorders) | 1 | NA
Dysgeusia (Nervous system disorders) | 1 | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Eye disorders - Other, specify (Eye disorders) | 1 | NA — Acute Posterior Vitreous Detachment OS
Fall (Injury, poisoning and procedural complications) | 1 | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | NA
Flu like symptoms (General disorders) | 1 | NA
General disorders and administration site conditions - Other, specify (General disorders) | 1 | NA — Cachetic
Hyperkalemia (Metabolism and nutrition disorders) | 1 | NA
Hypokalemia (Metabolism and nutrition disorders) | 1 | NA
Hypotension (Vascular disorders) | 1 | NA
Hypothyroidism (Endocrine disorders) | 1 | NA
INR increased (Investigations) | 1 | NA
Insomnia (Psychiatric disorders) | 1 | NA
Leukocytosis (Blood and lymphatic system disorders) | 1 | NA
Lipase increased (Investigations) | 1 | NA
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 | NA — Severe Protein Calorie Malnutrition
Multi-organ failure - (General disorders) | 1 | NA — failure to thrive
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | NA
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | NA — Tachypnea
Sepsis (Infections and infestations) | 1 | NA
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | NA — Scattered erythematous patches on trunk and abdomen
Skin infection (Infections and infestations) | 1 | NA
Small intestinal obstruction (Gastrointestinal disorders) | 1 | NA
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | NA
Thyroid stimulating hormone increased (Investigations) | 1 | NA
Weight gain (Investigations) | 1 | NA
Oral dysesthesia (Gastrointestinal disorders) | 1 | NA
Scleral disorder (Eye disorders) | 1 | NA
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT04057365/Prot_SAP_000.pdf